CLINICAL TRIAL: NCT01909050
Title: An In-vitro Gluten Challenge on the Immunologic Response in Celiac Disease.
Brief Title: Immune Response in Celiac Disease on In-vitro Gluten Challenge
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Leffler, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2012P000354
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Celiac Disease
Keywords: celiac disease; refractory celiac disease; gluten sensitivity
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Duodenal biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- refractory celiac disease
- well-controlled celiac disease
- uncontrolled celiac disease: either newly diagnosed with celiac disease or not on a gluten-free diet
- gluten-sensitivity
- disorders other than celiac disease.

SUMMARY:
The main purpose of this study is to see how cells taken from the lining of the intestine behave in the laboratory with exposure to gluten and other substances that act on the immune system. The cells lining the intestine of a person with celiac disease should be different than a person without celiac disease. The study doctors would like to see how the cells react after coming in contact with gluten and if substances that act on the immune system can prevent gluten related inflammation. Examples of these substances include steroids. The cells should produce chemicals of their own in response to the gluten. These other chemicals will be measured and the results compared between those with:

* celiac disease that does not respond to a gluten-free diet (refractory celiac disease)
* celiac disease which is controlled by a gluten-free diet
* uncontrolled celiac disease (either newly diagnosed with celiac disease or not on a gluten-free diet
* gluten-sensitivity
* disorders other than celiac disease.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the effect of in-vitro introduction of gluten on inflammatory response primarily Interferon-γ and other cytokines, such as IL-15, IL-18 and IL-21, in cultures obtained from small intestinal mucosal biopsy samples of subjects who underwent upper endoscopy.

Secondary goals include comparing the inflammatory response to immunosuppressants and cytokines after exposing the cultures obtained from small intestinal mucosal biopsies taken from RCD I subjects with intestinal mucosal biopsies taken from subjects with CeD controlled on a Gluten-Free Diet (GFD), uncontrolled CeD, Gluten sensitivity and Non-celiac Controls.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Undergoing a clinically indicated upper endoscopy

Exclusion Criteria:

* Anticoagulation or antiplatelet therapy
* Known active non-celiac intestinal inflammatory disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients undergoing a clinically indicated upper endoscopy at Beth Israel Deaconess Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
change in interferon gamma | 0, 6, and 24 hours
  in vitro culture stimulated with gluten

SECONDARY OUTCOMES:
change in interleukin-15 | 0, 6, and 24 hours
  in vitro culture stimulated with gluten
change in interleukin-18 | 0, 6, and 24 hours
  in vitro culture stimulated with gluten
change in interleukin-21 | 0, 6, and 24 hours
  in vitro culture stimulated with gluten

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Leffler, MD, MS, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States